CLINICAL TRIAL: NCT07401303
Title: The Effect of Full-time RDI on the Incidence of Major Adverse Intraoperative or Delayed Events and the Proportion of ESD Procedures With Prolonged Procedure Time: A Multicenter Prospective Randomized Controlled Trial
Brief Title: Full-time RDI for ESD: Impact on Major Adverse Events and Procedure Time
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, MD, PhD, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJ-ESD-RDI
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Early Gastric Cancer or Gastric Adenoma
Keywords: endoscopic submucosal dissection; ESD; red dichromatic imaging; RDI; bleeding; perforation
MeSH Terms: conditions — Stomach Neoplasms; Hemorrhage | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-time RDI (Experimental): Full-time Red Dichromatic Imaging (RDI) refers to the continuous application of RDI technology throughout the entire endoscopic submucosal dissection (ESD) procedure. This approach encompasses all procedural phases, including submucosal injection, circumferential mucosal incision, submucosal dissection, and post-resection wound management, with the aim of enhancing visualization of submucosal vessels and bleeding sources in real time to improve hemostasis, reduce complications, and increase procedural efficiency.
  Interventions: Procedure: ESD
- Full-time WLI (Active Comparator): Full-time White Light Imaging (WLI) refers to the continuous use of standard white light endoscopic imaging throughout the entire endoscopic submucosal dissection (ESD) procedure. This conventional approach involves relying solely on white light visualization during all stages of the procedure-including submucosal injection, mucosal incision, submucosal dissection, and post-resection wound assessment-without the aid of enhanced imaging modalities for vessel or bleeding source identification.
  Interventions: Procedure: ESD

INTERVENTIONS:
Procedure: ESD — Endoscopic Submucosal Dissection (ESD) is a minimally invasive endoscopic technique used to remove early-stage gastrointestinal tumors and precancerous lesions en bloc. Developed initially for the treatment of early gastric cancer, ESD allows for precise dissection of the submucosal layer beneath the lesion, enabling complete resection with clear margins while preserving the integrity of the surrounding tissue. This technique offers advantages over traditional endoscopic mucosal resection (EMR) by enabling the removal of larger and more complex lesions, reducing recurrence rates, and minimizing the need for invasive surgery.
  Other Names: Endoscopic Submucosal Dissection

SUMMARY:
Gastric cancer remains a major global health burden, ranking fifth in incidence worldwide and disproportionately affecting Asia, with China accounting for a significant share of cases and deaths. Early detection and minimally invasive treatment are critical to improving outcomes. Endoscopic submucosal dissection (ESD) is the preferred curative approach for early gastric cancer, enabling precise, en bloc tumor resection while preserving gastric function. However, ESD is technically complex, time-consuming, and associated with risks such as intraoperative and delayed bleeding and perforation. These complications limit its widespread adoption, particularly outside East Asia.

Traditional ESD relies on white light imaging (WLI), which offers limited visualization of submucosal vessels and bleeding sources. Red Dichromatic Imaging (RDI) is an emerging image-enhanced endoscopy technology that uses specific narrow-band wavelengths to enhance the contrast of deep blood vessels and active bleeding sites by exploiting hemoglobin's optical absorption characteristics. Preliminary studies indicate that RDI improves bleeding point identification, facilitates hemostasis, and reduces endoscopists' procedural stress. However, prior research applied RDI only intermittently during bleeding events, leaving its potential benefits throughout the entire ESD procedure unexplored.

The "full-time RDI" concept proposes continuous use of RDI during all ESD stages-including submucosal injection, mucosal incision, dissection, and wound management-to enhance visualization of high-risk vessels, improve layer differentiation, and potentially reduce adverse events and operation time. Despite promising retrospective data, robust prospective evidence from large randomized controlled trials is lacking.

This multicenter, prospective randomized controlled trial aims to evaluate whether full-course RDI reduces major intraoperative and delayed complications and decreases unexpectedly prolonged operation times compared to conventional WLI-guided ESD in early gastric cancer. Secondary endpoints include procedural efficiency, safety across lesion locations, and operator stress.

By rigorously assessing full-time RDI's clinical value, this study addresses an urgent unmet need to improve ESD safety and efficiency, potentially broadening its application and enhancing patient outcomes. The innovation lies in integrating continuous advanced imaging throughout ESD, representing a significant advancement in endoscopic oncology and minimally invasive gastric cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo ESD for an early gastric cancer (the indication for ESD under current guidelines)
* both genders aged 18-75 years
* no pretreatment (ESD, surgery, radiation therapy, or chemotherapy) performed on the stomach to be examined
* platelet count of >10×10^9/L and hemoglobin count of >8.0 g/L in blood tests performed in the 3 months before the ESD
* "antithrombotic drugs" have been withdrawn for the period recommended by current guidelines
* written consent provided at the patient's discretion

Exclusion Criteria:

* scheduled for hybrid ESD
* scheduled for ESD due to multiple lesions
* scheduled for treatment of lesions with residual recurrence
* presence of submucosal tumors
* unable to discontinue an antithrombotic drugs at the time of informed consent
* inherited or acquired coagulopathy likely to affect the risk of bleeding
* receiving maintenance dialysis
* deemed unsuitable for participation in this study by the principal investigator or other investigators
* unable to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of major intraoperative or delayed adverse events and/or ESD procedures with operation time exceeding the expected duration | From enrollment to the end of treatment at 4 weeks
  Major adverse events include use of hemostatic forceps for bleeding control, significant delayed bleeding, and perforation during or after ESD. Hemostatic forceps are used if bleeding persists after three electrocautery attempts or if the operator deems electrocautery insufficient. Delayed bleeding occurs mostly within 48 hours, marked by clinical signs needing hemostasis or transfusion, or >20 g/L hemoglobin drop. Perforation is diagnosed by visible gastric wall defects or post-ESD peritoneal irritation with free gas on imaging. Expected ESD time (min) = 2.384 × tumor size (mm) + 38.568 × location (1=upper third, 0=others) + 40.333 × ulcer presence (1=yes, 0=no). Procedures exceeding 110% of this time are analyzed by lesion and specimen size.

SECONDARY OUTCOMES:
Incidence of major intraoperative or delayed adverse events | From enrollment to the end of treatment at 4 weeks
  Major adverse events include use of hemostatic forceps for bleeding control, significant delayed bleeding, and perforation during or after ESD. Hemostatic forceps are applied before lesion removal and used until bleeding is fully controlled if: (1) bleeding persists after three electrocautery attempts; (2) the operator judges electrocautery insufficient; or (3) exposed vessels cannot be controlled by electrocautery. Use is allowed if either condition (2) or (3) applies, even without (1). Delayed bleeding usually occurs within 48 hours but can last up to 2 weeks, defined by clinical signs (hypotension, tachycardia, hematemesis, melena, hematochezia) requiring endoscopic hemostasis or transfusion, or hemoglobin drop >20 g/L. Intraoperative perforation is a visible gastric wall defect with exposed fat or peritoneal cavity; delayed perforation shows peritoneal irritation and free gas on postoperative imaging.
Incidence of ESD procedures exceeding 110% of the expected procedure time | Throughout the ESD procedure
  Expected operation time = 2.384 × tumor size (mm) + 38.568 × location + 40.333 × ulcer presence; where location is assigned 1 for tumors in the upper third of the stomach and 0 for tumors in the middle or lower third; ulcer presence is assigned 1 if ulcers are present and 0 if absent.
  An ESD procedure is considered to exceed 110% of the expected operation time if its actual duration surpasses the estimated time by more than 10%. Analyses can be performed separately based on the preoperative estimated lesion size and the size of the resected specimen.
Number of ESD procedures requiring hemostatic forceps for hemostasis | Throughout the ESD procedure
  The outcome measure reports the number of ESD procedures requiring hemostatic forceps for bleeding control. Procedures were counted as requiring hemostatic forceps if forceps were applied to achieve hemostasis during the procedure. The count ranges from zero (no procedures requiring forceps) to the total number of ESD procedures performed.
Number of hemostatic forceps uses during ESD | Throughout the ESD procedure
  The outcome measure reports the number of times hemostatic forceps were used during ESD. The count ranges from zero, indicating no use of hemostatic forceps, to the maximum number of uses recorded during the procedure. A higher count reflects more frequent use of hemostatic forceps for bleeding control during ESD.
Number of hemostatic interventions during the procedure (regardless of type) | Throughout the ESD procedure
  The outcome measure reports the number of hemostatic interventions performed during the procedure, regardless of the intervention type. The count ranges from zero, indicating no hemostatic intervention was required, to the maximum number of interventions recorded in a procedure. A higher count indicates more frequent hemostatic interventions to control bleeding during the procedure.
Number of spurting hemorrhages (Forrest classification Ia) | Throughout the ESD procedure
  The outcome measure reports the number of spurting hemorrhages classified as Forrest Ia observed during the procedure. The count ranges from zero, indicating no spurting hemorrhages, to the maximum number identified. A higher number reflects a greater severity of active arterial bleeding according to the Forrest classification.
Procedure time (minutes) and submucosal dissection time (minutes) | Throughout the ESD procedure
  Procedure time (minutes) is defined as the time from the start of mucosal incision to the complete removal of the lesion. Submucosal dissection time (minutes) is defined as the time from the completion of circumferential mucosal incision to the end of complete lesion removal. The outcome measures report time durations in minutes.
Dissection speed (mm²/min) | Throughout the ESD procedure
  The outcome measure reports dissection speed in mm²/min, which is calculated by dividing the specimen area (mm²) by the submucosal dissection time (minutes). Specimen area is determined using the elliptical formula: area (mm²) = longest diameter (mm) × shortest diameter (mm) × 0.25 × 3.14. Dissection speed ranges from zero (no tissue dissected per minute) to the maximum speed recorded. Higher values indicate faster dissection during the procedure.
Volume of submucosal injection solution used | Throughout the ESD procedure
  The outcome measure reports the volume of submucosal injection solution used, calculated as the initial prepared volume minus the remaining volume (measured in milliliters, ml). The volume ranges from zero, indicating no solution was used, to the maximum amount prepared. Greater volumes reflect higher usage of injection solution during the procedure.
Rates of en bloc resection | From enrollment to the end of treatment at 4 weeks
  En bloc resection is defined as the complete removal of the target lesion in a single piece without piecemeal resection. Participants are considered to have achieved this outcome if their lesions meet these criteria. Rates range from 0% (no participants achieving the outcome) to 100% (all participants achieving the outcome), with higher rates indicating better procedural success.
Rates of complete resection | From enrollment to the end of treatment at 4 weeks
  Complete resection is confirmed by histological examination showing negative horizontal and vertical margins. Participants are considered to have achieved this outcome if their lesions meet these criteria. Rates range from 0% (no participants achieving the outcome) to 100% (all participants achieving the outcome), with higher rates indicating better procedural success.
Rates of curative resection | From enrollment to the end of treatment at 4 weeks
  Curative resection is determined according to the Japanese Gastric Cancer Guidelines, classified as endoscopic cure categories A, C-1, and C-2.
  Participants are considered to have achieved this outcome if their lesions meet these criteria. Rates range from 0% (no participants achieving the outcome) to 100% (all participants achieving the outcome), with higher rates indicating better procedural success.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi, China